CLINICAL TRIAL: NCT00391612
Title: A Randomized, Double-blind Study to Evaluate the Safety and Effectiveness of the Exhale® Drug-Eluting Stent in Homogeneous Emphysema Subjects With Severe Hyperinflation
Brief Title: EASE Trial: Exhale Airway Stents for Emphysema
Acronym: EASE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Broncus Technologies (Industry)
Responsible Party: Nancy Isaac, Senior Vice President, Clinical and Regulatory Affairs and Quality Assurance, Broncus Technologies, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol 30
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Emphysema
Keywords: COPD (Chronic Obstructive Pulmonary Disease); Emphysema; Hyperinflation; Minimally Invasive
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 2 (Sham Comparator): subject receives optimal medical management, supervised pulmonary rehabilitation therapy and undergoes bronchoscopy but no stents are placed
  Interventions: Device: Sham control
- 1 (Experimental): subject receives optimal medical management, supervised pulmonary rehabilitation therapy and undergoes bronchoscopy during which up to six Exhale drug-eluting stents are placed in the lungs
  Interventions: Device: Exhale® Drug-Eluting Stent

INTERVENTIONS:
Device: Exhale® Drug-Eluting Stent — Bronchoscopic procedure in which up to six Exhale Drug-Eluting Stents are placed in the lungs; total procedure time is 1 to 2 hours
  Arms: 1
Device: Sham control — 5-10 minute bronchoscopic procedure in which the lungs are examined and a bronchial lavage is performed; the bronchoscope is then retracted to a point above the carina and below the vocal folds for the remained of the time; total procedure time is about 1-2 hours
  Arms: 2

SUMMARY:
This is an international clinical research study evaluating the safety and effectiveness of a new procedure called airway bypass. The goal of this research is to see if airway bypass can relieve hyperinflation (overfilling) of the lungs, thereby improving lung function and reducing shortness of breath in patients with severe homogeneous (diffuse) emphysema. "EASE" stands for Exhale Airway Stents for Emphysema.

DETAILED DESCRIPTION:
Over 3 million people in the United States and tens of millions more throughout the world live with emphysema, a chronic, progressive, irreversible disease of the lungs. The hallmark of emphysema is hyperinflation of the lungs -- air is trapped in the lungs and cannot escape, causing the lungs to become larger and larger. This makes it difficult to breathe and dyspnea (shortness of breath) is the result.

The airway bypass procedure is performed using a bronchoscope with the patient under anesthesia. Very small passageways are created between the damaged lung tissue and the larger breathing passages (airways). Small stents are inserted to keep the new pathways from closing. These pathways could potentially provide a way for the trapped air to escape when the patient exhales. If the amount of air trapped in the lungs is reduced then it should be easier for the person to breathe.

The EASE study will compare the effects of Exhale Drug-Eluting Stents in patients to a sham-control group of patients who do not receive the stents. Two out of three (2/3) of the participants in the trial will be in the airway bypass group, or "treatment" group. Participants in the treatment group will undergo the airway bypass procedure with up to six drug-eluting stents implanted in their lungs, creating the passageways for the trapped air to escape. A smaller group - one out of three (1/3) participants - will be the "control" group. The control group will have bronchoscopy, but passages will not be made and stents will not be implanted.

Participants will need to return to the study center four times during the year for follow-up visits and tests. All participants will be told which group they were in when they come back for a follow-up visit one year after the procedure. Participants in the control group will be finished with the trial after one year. Participants in the treatment group will have a follow-up visit once a year for the next four years to monitor the longer term effects of the airway bypass procedure. This is why the end date of the trial is listed as 2012.

ELIGIBILITY:
Inclusion Criteria:

1. High resolution computed tomography (CT) scan evidence of homogeneous emphysema.
2. Stopped smoking at least 8 weeks before entering the trial.
3. Post-bronchodilator RV/TLC ≥ 0.65.
4. Post-bronchodilator Forced Expiratory Volume (FEV1) ≤ 50% or FEV1 < 1 liter.
5. Marked dyspnea, scoring ≥ 2 on the modified Medical Research Council scale of 0-4.
6. Patient has undergone supervised pulmonary rehabilitation of 16-20 sessions over 6-10 weeks.

Exclusion Criteria:

1. Change in FEV1 > 20% pre- and post- bronchodilator measurements or > 200 ml if post-bronchodilator FEV1 < 1 liter.
2. Respiratory infections requiring 3 or more hospitalizations in past year.
3. Inability to walk > 140 meters (150 yards) in 6 minutes.
4. Previous lung volume reduction surgery (LVRS) or lobectomy.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 6 months
modified Medical Research Council (mMRC) score (breathlessness) | 6 months

SECONDARY OUTCOMES:
Residual Volume/Total Lung Capacity (RV/TLC) | 6 months
Forced Vital Capacity (FVC) | 6 months
modified Medical Research Council Dyspnea Scale (mMRC) | 6 months
Forced Expiratory Volume in 1 second (FEV1) | 6 months
St. George's Respiratory Questionnaire (SGRQ) | 6 months
6-minute walk (6MW) | 6 months
Cycle Ergometry | 6 months
Note: Residual Volume/Total Lung Capacity (RV/TLC) will be analyzed for superiority. All other secondary endpoints will be analyzed for informational purposes. | 6 months
Residual Volume (RV) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel D. Cooper, MD, FACS, FRCS, Principal Investigator; Gerhard W. Sybrecht, Prof. Dr. med., Principal Investigator — Universitätskliniken des Saarlandes
Locations (37):
- United States (26):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - UCSF-Fresno, Fresno, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Emory Healthcare, Atlanta, Georgia
  - Peoria Pulmonary Associates, LTD, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Chicago Chest Center at Central DuPage Hospital, Winfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Topeka Pulmonary/Veritas Clinical Specialties, LTD, Topeka, Kansas
  - Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital & Medical Center, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - International Heart Institute of Montana Foundation, Missoula, Montana
  - New York Methodist Hospital, Brooklyn, New York
  - New York University - Bellevue Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- The Alfred Hospital, Melbourne, Victoria, Australia
- Otto Wagner Hospital, Vienna, Austria
- Santa Casa Hospital, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Hopital Laval, Québec, Quebec
- Universitatsklinik des Saarlandes, Homburg, Saarland, Germany
- Mater Misericordiae University Hospital, Dublin, Ireland
- University Medical Center, Groningen, Groningen, Netherlands
- Fundación Jiménez Díaz, Madrid, Spain
- United Kingdom (2):
  - Papworth Hospital, Cambridge
  - The Royal Brompton Hospital, London

REFERENCES:
- [Background] Lausberg HF, Chino K, Patterson GA, Meyers BF, Toeniskoetter PD, Cooper JD. Bronchial fenestration improves expiratory flow in emphysematous human lungs. Ann Thorac Surg. 2003 Feb;75(2):393-7; discussion 398. doi: 10.1016/s0003-4975(02)04553-8. PMID 12607646
- [Background] Rendina EA, De Giacomo T, Venuta F, Coloni GF, Meyers BF, Patterson GA, Cooper JD. Feasibility and safety of the airway bypass procedure for patients with emphysema. J Thorac Cardiovasc Surg. 2003 Jun;125(6):1294-9. doi: 10.1016/s0022-5223(02)73243-1. PMID 12830047
- [Background] Choong CK, Haddad FJ, Gee EY, Cooper JD. Feasibility and safety of airway bypass stent placement and influence of topical mitomycin C on stent patency. J Thorac Cardiovasc Surg. 2005 Mar;129(3):632-8. doi: 10.1016/j.jtcvs.2004.07.062. PMID 15746748
- [Background] Choong CK, Phan L, Massetti P, Haddad FJ, Martinez C, Roschak E, Cooper JD. Prolongation of patency of airway bypass stents with use of drug-eluting stents. J Thorac Cardiovasc Surg. 2006 Jan;131(1):60-4. doi: 10.1016/j.jtcvs.2005.07.057. Epub 2005 Dec 5. PMID 16399295
- [Background] Terry PB, Traystman RJ, Newball HH, Batra G, Menkes HA. Collateral ventilation in man. N Engl J Med. 1978 Jan 5;298(1):10-5. doi: 10.1056/NEJM197801052980103. PMID 618444
- [Background] Macklem PT. Collateral ventilation. N Engl J Med. 1978 Jan 5;298(1):49-50. doi: 10.1056/NEJM197801052980112. No abstract available. PMID 618452
- [Background] Choong CK, Macklem PT, Pierce JA, Lefrak SS, Woods JC, Conradi MS, Yablonskiy DA, Hogg JC, Chino K, Cooper JD. Transpleural ventilation of explanted human lungs. Thorax. 2007 Jul;62(7):623-30. doi: 10.1136/thx.2005.053256. Epub 2007 Apr 5. PMID 17412776
- [Background] Cardoso PF, Snell GI, Hopkins P, Sybrecht GW, Stamatis G, Ng AW, Eng P. Clinical application of airway bypass with paclitaxel-eluting stents: early results. J Thorac Cardiovasc Surg. 2007 Oct;134(4):974-81. doi: 10.1016/j.jtcvs.2007.05.040. Epub 2007 Aug 20. PMID 17903516
- [Derived] Shah PL, Slebos DJ, Cardoso PF, Cetti E, Voelker K, Levine B, Russell ME, Goldin J, Brown M, Cooper JD, Sybrecht GW; EASE trial study group. Bronchoscopic lung-volume reduction with Exhale airway stents for emphysema (EASE trial): randomised, sham-controlled, multicentre trial. Lancet. 2011 Sep 10;378(9795):997-1005. doi: 10.1016/S0140-6736(11)61050-7. PMID 21907863
- [Derived] Shah PL, Slebos DJ, Cardoso PF, Cetti EJ, Sybrecht GW, Cooper JD. Design of the exhale airway stents for emphysema (EASE) trial: an endoscopic procedure for reducing hyperinflation. BMC Pulm Med. 2011 Jan 7;11:1. doi: 10.1186/1471-2466-11-1. PMID 21214899
- See also: Broncus Technologies, Inc., corporate web page. — http://www.broncus.com
- See also: American Lung Association — http://www.lungusa.org